CLINICAL TRIAL: NCT05510024
Title: Radiofrequency Ablation of Bilateral Inferior Turbinate Followed by Subcutaneous Immunotherapy Trial for Severe House Dust Mite-sensitized Allergic Rhinitis
Brief Title: Radiofrequency Ablation of Bilateral Inferior Turbinate Followed by Subcutaneous Immunotherapy Trial
Acronym: RABIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Huabin Li, Chief of Department of Allergy, Eye & ENT Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RABIT-2022
Record Dates: First submitted 2022-06-08; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Allergic Rhinitis Due to House Dust Mite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors who were involved in outcome measurements will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency ablation of bilateral inferior turbinate followed by subcutaneous Immunotherapy (Experimental): Radiofrequency ablation of bilateral inferior turbinate followed by subcutaneous Immunotherapy will be conducted in participants with severe house dust mite-sensitized allergic rhinitis.
  Interventions: Procedure: Radiofrequency ablation of bilateral inferior turbinate followed by subcutaneous immunotherapy
- Subcutaneous Immunotherapy (SCIT) (Active Comparator): Allergen-specific subcutaneous Immunotherapy will be conducted in participants with severe house dust mite-sensitized allergic rhinitis.
  Interventions: Procedure: SCIT

INTERVENTIONS:
Procedure: Radiofrequency ablation of bilateral inferior turbinate followed by subcutaneous immunotherapy — The regulation and monitoring of the entire soft-coagulation process are conducted via the radiofrequency generator under endoscopic guidance. Lateral out-fracture of the inferior turbinate is performed if necessary. One month after surgery, allergen immunotherapy will be conducted. Standardized Dp allergen extracts (Alutard SQ, ALK-Abell'o) were used for SCIT. According to the manufacturer's instructions, the build up phase was carried out with weekly injections of volumes of 0.2, 0.4, and 0.8 mL in the first 3 vials (nos. 1 to 3) and 0.1, 0.2, 0.4, 0.8, and 1.0 mL in vial no. 4, reaching the maintenance dose, 100,000 standardized quality units. The specialist adjusted the dose according to the patient's therapeutic response, and the cumulative allergen dose for each patient was the maximal tolerable injected dose. Then, the maintenance dose was given with an injection interval of 6±2 weeks according to the manufacturer's recommendations.
  Arms: Radiofrequency ablation of bilateral inferior turbinate followed by subcutaneous Immunotherapy
Procedure: SCIT — Allergen immunotherapy will be conducted. Standardized Dp allergen extracts (Alutard SQ, ALK-Abell'o) were used for SCIT. According to the manufacturer's instructions, the build up phase was carried out with weekly injections of volumes of 0.2, 0.4, and 0.8 mL in the first 3 vials (nos. 1 to 3) and 0.1, 0.2, 0.4, 0.8, and 1.0 mL in vial no. 4, reaching the maintenance dose, 100,000 standardized quality units. The specialist adjusted the dose according to the patient's therapeutic response, and the cumulative allergen dose for each patient was the maximal tolerable injected dose. Then, the maintenance dose was given with an injection interval of 6±2 weeks according to the manufacturer's recommendations.
  Arms: Subcutaneous Immunotherapy (SCIT)

SUMMARY:
Allergic rhinitis (AR) is a global health issue adversely impacting the quality of life (QoL) of affected individuals and exerting a huge public health burden. Allergen immunotherapy (AIT) has been shown to be effective in the treatment of not only the symptoms, but also the underlying causes of the disease. Moreover, AIT has a preventative role against new sensitizations and development of asthma in AR patients. Hence AIT is recommended as an integrated part of an allergy management strategy in the treatment of AR. Over the development of one century, AIT has been delivered by various routes. Among them, subcutaneous immunotherapy (SCIT) has been currently widely used in clinical practice.

House dust mite (HDM) has been reported to be the most common sensitizing allergen in China. Nasal obstruction is the common complaint in HDM-sensitized AR and prompts patients to seek medical help. It has been proved that HDM-SCIT showed favourable efficacy in treating persistent AR. However, HDM-SCIT recommends 3 years of subcutaneous injection and requires good adherence to guarantee the efficacy. Later onset of nasal obstruction alleviation might reduce the adherence of HDM-SCIT.

Radiofrequency ablation of bilateral inferior turbinate can relieve nasal obstruction within a short time after operation. It is hypothesized that, in HDM-AR patients with severe nasal obstruction, bilateral inferior turbinate surgery followed by HDM-SCIT will obtain quick-onset of good nasal ventilation and improve AIT adherence.

The overall objective of the proposed randomized controlled trial is to test whether radiofrequency ablation of bilateral inferior turbinate followed by subcutaneous immunotherapy will improve nasal obstruction among patients with house dust mite sensitized allergic rhinitis (HDM-AR) compared to subcutaneous immunotherapy (SCIT) only during the 4-month build-up phase as well as the 36-month full phase of SCIT.

DETAILED DESCRIPTION:
The overall objective of the proposed randomized controlled trial is to test whether radiofrequency ablation of bilateral inferior turbinate followed by subcutaneous immunotherapy will improve nasal obstruction among patients with house dust mite sensitized allergic rhinitis (HDM-AR) compared to subcutaneous immunotherapy (SCIT) only during the 4-month build-up phase as well as the 36-month full phase of SCIT.

Specifically, the investigator propose to conduct a multicentre randomized trial to achieve the following specific aims:

1. To test whether radiofrequency ablation of bilateral inferior turbinate plus subcutaneous immunotherapy (RABIT) will improve nasal obstruction over a 4-month build-up phase of SCIT compared to subcutaneous immunotherapy (SCIT) only among patients with HDM-AR in China;
2. To test whether RABIT will improve each nasal symptom of AR, including sneezing, nasal itching, rhinorrhea and nasal congestion over the 36-month full phase of SCIT compared to SCIT only among patients with HDM-AR in China;
3. To evaluate whether RABIT will improve health-related quality of life (HRQoL) compared to SCIT only among patients with HDM-AR in China;
4. To estimate the cost-effectiveness of RABIT compared to SCIT only in China.
5. To test whether RABIT will decrease the risk of incidence of asthma and reduce new sensitizations compared to SCIT only in China.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 60 years
* at least 2-year history of physician-diagnosed HDM-AR, with positive skin prick test to house dust mite and/or positive serum antigen-specific IgE
* nasal congestion score ≥7, severe inferior turbinate hypertrophy (no visible of middle turbinate)
* no oral steroids for 4 weeks prior to treatment
* no intranasal steroids and/or antihistamines for 2 weeks prior to recruitment

Exclusion Criteria:

* symptomatic seasonal AR
* any respiratory infection within the previous 4 weeks prior to recruitment
* chronic rhinosinusitis with or without nasal polyps, nasal septum deviation, cleft lip and/or palate, autoimmune disorders, malignant tumor, immune deficiency disease, tuberculosis, cardiac dysfunction, uncontrolled asthma, beta blocker in taker, other severe systemic disease
* pregnancy or breastfeeding females
* those who had previously received AIT or nasal surgery within one month or those who participated other clinical trials within 3 months prior to recruitment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 392 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in nasal congestion score (NCS) | baseline (Visit 0), one month after surgery (Visit 1, before first injection in SCIT), end of build up phase (Visit2, up to four months after first injection), up to 12 months (Visit 3), up to 24 months (Visit 4), up to 36 months (Visit5)
  Nasal congestion is graded on a visual analog scale score (0, none; 10, severe). (1) Phase I: change in NCS during the 4-month build-up phase of SCIT between the intervention and control groups (2) Phase II: differences in NCS over the 36-month full phase of subcutaneous immunotherapy (SCIT) between the intervention and control groups.

SECONDARY OUTCOMES:
TNSS | baseline (Visit 0), one month after surgery (Visit 1, before first injection in SCIT), end of build up phase (Visit2, up to four months after first injection), up to 12 months (Visit 3), up to 24 months (Visit 4), up to 36 months (Visit5)
  total nasal symptoms score including nasal congestion, rhinorrhea, itching and sneezing
total combined score (TCS) | baseline (Visit 0), one month after surgery (Visit 1, before first injection in SCIT), end of build up phase (Visit2, up to four months after first injection), up to 12 months (Visit 3), up to 24 months (Visit 4), up to 36 months (Visit5)
  Total combined score (TCS) is calculated as the combined score of average scores of six nasal/conjunctivitis symptoms (rhinorrhea, nasal congestion, nasal itching, sneezing, gritty eyes, and watery eyes) and the rescue medication score (RMS), ranging from 0 to 6 (0, none; 6, severe).
Rescue medication score | baseline (Visit 0), one month after surgery (Visit 1, before first injection in SCIT), end of build up phase (Visit2, up to four months after first injection), up to 12 months (Visit 3), up to 24 months (Visit 4), up to 36 months (Visit5)
  The need for rescue medication was assessed throughout the treatment as rescue medication score (RMS), ranging from 0 to 3 as follows: 0 = no use of rescue medication, 1 = use of oral and/or topical non-sedative H1 antihistamines, 2 = use of intranasal corticosteroids with/without H1 antihistamines, and 3 = use of oral corticosteroids with/without intranasal corticosteroids, with/without H1 antihistamines.
Health-related quality of life | baseline (Visit 0), one month after surgery (Visit 1, before first injection in SCIT), end of build up phase (Visit2, up to four months after first injection), up to 12 months (Visit 3), up to 24 months (Visit 4), up to 36 months (Visit5)
  The rhinoconjunctivitis quality of life questionnaire (RQLQ) consisted of seven domains with a total of 28 questions. And the score was recorded at each visit to evaluate the quality of life.
Number of patients who achieve target maintenance dose | end of build up phase (Visit2, up to four months after first injection)
  Number of patients who achieve target maintenance dose
Incidence rate of asthma and new sensitizations | baseline (Visit 0), up to 12 months (Visit 3), up to 24 months (Visit 4), up to 36 months (Visit5)
  Incidence rate of asthma on those who did not have asthma at baseline
cost effectiveness ratio | baseline (Visit 0), up to 36 months (Visit5)
  Primary incremental cost effectiveness ratio (ICER) measures will be cost per % change in nasal congestion score
adverse events | baseline (Visit 0), one month after surgery (Visit 1, before first injection in SCIT), end of build up phase (Visit2, up to four months after first injection), up to 12 months (Visit 3), up to 24 months (Visit 4), up to 36 months (Visit5)
  Safety was evaluated by the occurrence and severity of adverse events (AEs) and the casual relationship between AEs and the experimental drug. All AEs will be categorized as mild (no impact on the activities of daily living), moderate (decreased or affected performance of the activities of daily living) or severe (an inability to perform the activities of daily living or death).

CONTACTS AND LOCATIONS:
Overall Officials: Huabin Li, Principal Investigator — Eye & ENT Hospital of Fudan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brozek JL, Bousquet J, Agache I, Agarwal A, Bachert C, Bosnic-Anticevich S, Brignardello-Petersen R, Canonica GW, Casale T, Chavannes NH, Correia de Sousa J, Cruz AA, Cuello-Garcia CA, Demoly P, Dykewicz M, Etxeandia-Ikobaltzeta I, Florez ID, Fokkens W, Fonseca J, Hellings PW, Klimek L, Kowalski S, Kuna P, Laisaar KT, Larenas-Linnemann DE, Lodrup Carlsen KC, Manning PJ, Meltzer E, Mullol J, Muraro A, O'Hehir R, Ohta K, Panzner P, Papadopoulos N, Park HS, Passalacqua G, Pawankar R, Price D, Riva JJ, Roldan Y, Ryan D, Sadeghirad B, Samolinski B, Schmid-Grendelmeier P, Sheikh A, Togias A, Valero A, Valiulis A, Valovirta E, Ventresca M, Wallace D, Waserman S, Wickman M, Wiercioch W, Yepes-Nunez JJ, Zhang L, Zhang Y, Zidarn M, Zuberbier T, Schunemann HJ. Allergic Rhinitis and its Impact on Asthma (ARIA) guidelines-2016 revision. J Allergy Clin Immunol. 2017 Oct;140(4):950-958. doi: 10.1016/j.jaci.2017.03.050. Epub 2017 Jun 8. PMID 28602936
- [Background] Durham SR, Penagos M. Sublingual or subcutaneous immunotherapy for allergic rhinitis? J Allergy Clin Immunol. 2016 Feb;137(2):339-349.e10. doi: 10.1016/j.jaci.2015.12.1298. PMID 26853126
- [Background] Lou H, Ma S, Zhao Y, Cao F, He F, Liu Z, Bousquet J, Wang C, Zhang L, Bachert C. Sensitization patterns and minimum screening panels for aeroallergens in self-reported allergic rhinitis in China. Sci Rep. 2017 Aug 24;7(1):9286. doi: 10.1038/s41598-017-10111-9. PMID 28839248
- [Background] Ciprandi G, Cirillo I, Vizzaccaro A, Tosca M, Passalacqua G, Pallestrini E, Canonica GW. Seasonal and perennial allergic rhinitis: is this classification adherent to real life? Allergy. 2005 Jul;60(7):882-7. doi: 10.1111/j.1398-9995.2005.00602.x. PMID 15932377
- [Background] Karakoc-Aydiner E, Eifan AO, Baris S, Gunay E, Akturk E, Akkoc T, Bahceciler NN, Barlan IB. Long-Term Effect of Sublingual and Subcutaneous Immunotherapy in Dust Mite-Allergic Children With Asthma/Rhinitis: A 3-Year Prospective Randomized Controlled Trial. J Investig Allergol Clin Immunol. 2015;25(5):334-42. PMID 26727762
- [Background] Sahin E, Dizdar D, Dinc ME, Cirik AA. Long-term effects of allergen-specific subcutaneous immunotherapy for house dust mite induced allergic rhinitis. J Laryngol Otol. 2017 Nov;131(11):997-1001. doi: 10.1017/S0022215117002110. Epub 2017 Oct 17. PMID 29037263
- [Background] Tabar AI, Arroabarren E, Echechipia S, Garcia BE, Martin S, Alvarez-Puebla MJ. Three years of specific immunotherapy may be sufficient in house dust mite respiratory allergy. J Allergy Clin Immunol. 2011 Jan;127(1):57-63, 63.e1-3. doi: 10.1016/j.jaci.2010.10.025. PMID 21211641
- [Background] Sohn MH. Efficacy and Safety of Subcutaneous Allergen Immunotherapy for Allergic Rhinitis. Allergy Asthma Immunol Res. 2018 Jan;10(1):1-3. doi: 10.4168/aair.2018.10.1.1. No abstract available. PMID 29178670